CLINICAL TRIAL: NCT01037647
Title: VLDL-triglyceride Kinetics and -Metabolism in the Post Absorptive State and During Hyperinsulinemia in Type 2 Diabetes
Brief Title: VLDL-triglyceride Kinetics in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: The Danish Medical Research Council (Other); The Novo Nordic Foundation (Other); The Danish Diabetes Association (Other)
Responsible Party: Sponsor
Other Study IDs: 20070028
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2011-11-07 (Estimated); Status verified 2011-11

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Diabetic dyslipidemia; VLDL-TG kinetics; VLDL-TG metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples Subcutaneous adipose tissue biopsies Muscle biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 2 diabetic men: Men with type 2 diabetes
  Interventions: Other: Hyperinsulinemic euglycemic glucose clamp
- Healthy men: Healthy men
  Interventions: Other: Hyperinsulinemic euglycemic glucose clamp

INTERVENTIONS:
Other: Hyperinsulinemic euglycemic glucose clamp — Hyperinsulinemic euglycemic glucose clamp, duration 5 hours, plasma glucose 5 mmol/l, insulin dosage 1,0 mU•kg FFM/min, human insulin (Actrapid; Novo Nordisk A/S).

SUMMARY:
Type 2 diabetes is associated with diabetic dyslipidemia, which is a major risk factor for coronary heart disease. Triglycerides (TG) and cholesterol are transported in the system of lipoproteins, and the metabolism of these lipids in plasma is closely interrelated. Evidence suggests that increased concentration of very low-density lipoprotein triglyceride (VLDL-TG) is a central pathophysiological feature of the lipid and lipoprotein abnormalities in diabetic dyslipidemia.

The objective of this study was to investigate VLDL-TG kinetics and aspects of peripheral VLDL-TG metabolism, i.e. to what extent VLDL-TG associated fatty acids (FA) are oxidized or deposited in regional adipose tissue, in subjects with type 2 diabetes and healthy controls in the postabsorptive state and during acute hyperinsulinemia using ex-vivo labeled VLDL-TG tracers.

ELIGIBILITY:
Inclusion Criteria:

Exclusion Criteria:

* Known disease except type 2 diabetes (type 2 diabetic subjects)
* Smoking
* Alcohol abuse
* Prescription medication expect oral antidiabetics (type 2 diabetic subjects)

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 11 men with type diabetes and 11 healthy men, matched for age and BMI.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2008-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
VLDL-TG production and clearance rates

SECONDARY OUTCOMES:
VLDL-TG oxidation
VLDL-TG subcutaneous adipose tissue storage

CONTACTS AND LOCATIONS:
Overall Officials: Søren Nielsen, DMSc, Principal Investigator — Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Denmark
Locations (1):
- Medical department M (Endocrinology and Diabetes), Aarhus University Hospital, Aarhus, DK, Denmark

REFERENCES:
- [Derived] Andersen IR, Sondergaard E, Sorensen LP, Nellemann B, Gormsen LC, Jensen MD, Nielsen S. Increased VLDL-TG Fatty Acid Storage in Skeletal Muscle in Men With Type 2 Diabetes. J Clin Endocrinol Metab. 2017 Mar 1;102(3):831-839. doi: 10.1210/jc.2016-2979. PMID 27898284
- [Derived] Sorensen LP, Andersen IR, Sondergaard E, Gormsen LC, Schmitz O, Christiansen JS, Nielsen S. Basal and insulin mediated VLDL-triglyceride kinetics in type 2 diabetic men. Diabetes. 2011 Jan;60(1):88-96. doi: 10.2337/db10-0564. Epub 2010 Sep 21. PMID 20858686